CLINICAL TRIAL: NCT06731322
Title: Gut, Inflammation and Nutrition in Adult Patients After Fontan Operation (GIN-Fontan Study)
Brief Title: Gut, Inflammation and Nutrition in Adult Patients After Fontan Operation
Acronym: GIN-Fontan
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Nejc Pavsic, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: 20240021
Record Dates: First submitted 2024-12-04; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Fontan Circulation; Fontan Procedure
Keywords: Fontan procedure, gut, inflammation, nutrition
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood sample for additional serum biomarker assesment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fontan operation group: Adults (>18 years old) after Fontan operation and without active protein-losing enteropathy
- Control group: Adults (>18 years old) with simple congenital heart defects without significant residual lesions or comorbidities

SUMMARY:
This observational case-control study aims to investigate intestinal barrier dysfunction, systemic inflammation, and nutritional status in adult patients after Fontan operation. Fontan operation, a palliative intervention for complex congenital heart defects, leads to an elevated systemic venous pressure, contributing to systemic complications, including gastrointestinal disturbances and liver disease. While protein-losing enteropathy (PLE) is a known complication, this study focuses on patients without PLE to assess less-studied effects on the gastrointestinal system.

The elevated systemic venous pressure in adult patients after Fontan operation may impair the protective and absorptive functions of the gastrointestinal tract. This dysfunction allows bacterial endotoxins to enter the bloodstream, triggering systemic inflammation, which can worsen heart failure, cause malnutrition, and lead to cachexia. Although these outcomes are established in acquired heart failure, there is a lack of studies specifically examining the gastrointestinal consequences in adult patients after Fontan operation without PLE.

In this study, adult Fontan patients without PLE will be compared to a control group of patients with simple congenital heart defects and normal systemic venous pressure. The study will evaluate intestinal barrier dysfunction, systemic inflammatory responses, and malnutrition through several methods: serum biomarkers (I-FABP, LBP, TNF-α, IL-6, etc.), nutritional assessment including body composition assessment using bioelectrical impedance analysis and measurements of serum microelements, echocardiography, and abdominal ultrasound with liver elastography.

The findings of the study will help elucidate the connection between intestinal barrier dysfunction, inflammation, and nutritional status in adult patients after Fontan operation, aiming to improve long-term outcomes for this unique patient population.

DETAILED DESCRIPTION:
Clinical studies in patients with acquired heart disease and heart failure have shown that elevated systemic venous pressure is associated with significant venous congestion of the gastrointestinal tract and impairment of its protective and absorptive functions. The consequence of an impaired intestinal barrier is the entry of toxins (lipopolysaccharide or endotoxin), intestinal bacteria, or their metabolites into the bloodstream. In patients with decompensated heart failure, significantly higher levels of endotoxin were recorded, which were shown to decrease following treatment with diuretics. The translocation of bacterial toxins and metabolites across has been proven to trigger a systemic inflammatory response, which is considered a major factor in the progression of heart failure. Additionally, intestinal barrier dysfunction and systemic inflammatory response can lead to malnutrition and the development of cachexia, which is a poor prognostic factor in patients with heart failure.

Adult patients after Fontan operation represent a specific group of patients with congenital heart disease that is characterized by with long-term systemic venous pressure elevation. The Fontan procedure is a multistage palliative surgical intervention performed in patients with complex congenital heart defects where a bi-ventricular repair is not possible. In patients after Fontan operation, systemic venous blood from both inferior and superior venae cavae is surgically redirected into the pulmonary artery. The systemic venous circulation thus functions without an active pump (the right ventricle), so the flow to the pulmonary artery is passive. The pathophysiological consequence of establishing Fontan circulation is an elevated systemic venous pressure. Based on invasive hemodynamic studies the systemic venous pressure in patients after Fontan operation averages around 14 mmHg, which is approximately 3-4 times higher than normal systemic venous pressure (3-5 mmHg).

Patients after the Fontan operation experience numerous systemic complications and have a known reduced life expectancy. The most well-known and studied gastrointestinal consequences are liver damage with hepatopathy and the development of cirrhosis (Fontan-associated liver disease, FALD) and protein-losing enteropathy (PLE). Protein-losing enteropathy is recorded in 3-18% of patients after Fontan operation, and its occurrence is associated with elevated systemic venous pressure, disturbances in lymphatic circulation, and systemic inflammation.

The impact of the Fontan operation and its hemodynamic consequences on the protective and absorptive functions of the gastrointestinal tract in patients without signs of protein-losing enteropathy is unknown. Pathophysiologically, adult patients after Fontan operation have several factors that may contribute to impaired intestinal function. In addition to intestinal congestion due to elevated systemic venous pressure, reduced cardiac output may further contribute to impairment by leading to hypoperfusion and intestinal ischemia. Some patients after Fontan operation also have a surgical connection ("fenestration") that leads to a right-to-left cardiac shunt, hypoxemia, and cyanosis, which may further worsen intestinal blood flow.

Studies on intestinal barrier dysfunction in adult patients after Fontan operation who do not have protein-losing enteropathy are not available. A previous study on a group of patients with various congenital heart defects demonstrated intestinal barrier dysfunction with higher serum levels of bacterial endotoxin compared to healthy controls. These levels were higher in patients with concomitant signs of heart failure. Furthermore, patients with congenital heart defects had significantly elevated biomarkers of the systemic inflammatory response (tumour necrosis factor-alpha (TNFα) and interleukin-6 (IL-6)). Dysbiosis of intestinal bacteria, characterized by a pathologically altered composition of the gut microbiota, and a systemic inflammatory response with elevated levels of TNFα and IL-6, have also previously been demonstrated in patients after Fontan operation.

Additionally, changes in body composition, particularly pronounced myopenia, have been documented in patients after Fontan operation. However, studies on nutritional disorders in these patients are not available. Based on research in patients with acquired heart failure, intestinal barrier dysfunction and systemic inflammatory response lead to malnutrition and the development of cachexia.

Study Protocol

The study is designed as an observational case-control study. The investigators will include adult patients (older than 18 years) who have undergone Fontan operation and are followed up in the Adult Congenital Heart Disease Clinic at the Clinical Department of Cardiology, University Medical Centre Ljubljana. Patients with known active protein-losing enteropathy will be excluded. The control group will consist of patients who have undergone surgical or percutaneous repair of simple congenital heart defects (atrial or ventricular septal defects). Control patients will be without clinical signs of heart failure and with normal systemic venous pressure as assessed by ultrasound.

Methods

1. Laboratory Parameters

   Blood samples will be taken from both patients and controls to measure:

   Biomarkers of intestinal barrier dysfunction:

   I-FABP (Intestinal Fatty Acid-Binding Protein) - a marker of enterocyte damage. LBP (Lipopolysaccharide Binding Protein) - an indicator of serum bacterial endotoxin levels.

   Biomarkers of systemic inflammatory response:

   TNF-alpha (Tumor Necrosis Factor-α) IL-6 (Interleukin 6) IL-1B (Interleukin 1B) sCD14 (soluble CD14 protein receptor) hsCRP (high-sensitivity C-Reactive Protein)

   Micronutrients and vitamins:

   Calcium, Phosphate, Magnesium, Iron, Selenium, Folic Acid, Vitamin B12, Vitamin A, Vitamin E, Vitamin D, Folic acid
2. Nutritional Assessment Each participant will be evaluated by a clinical dietitian who will conduct a nutritional history and status examination. Nutritional disorders will be screened using the GLIM method, which includes nutritional status assessment with the MUST questionnaire and body composition assessment using bioelectrical impedance analysis.

   For further nutritional assessment, three clinical scoring systems will be used:

   GNRI (Geriatric Nutritional Risk Index) PNI (Prognostic nutritional index) CONUT (Controlling Nutritional Status)
3. Abdominal Ultrasound and Elastography Abdominal ultrasound will be performed to assess the morphology of the liver and signs of portal hypertension. Liver elastography will also be performed using two methods: FibroScan and shear wave elastography. Liver elastography will be used to non-invasively estimate systemic venous pressure (Fontan circulation pressure) as previously described.
4. Echocardiography Echocardiography will evaluate the function of the systemic ventricle, atrioventricular, and semilunar valves. Both qualitative and quantitative parameters will be used
5. Cardiopulmonary Exercise Testing This test will be performed on all patients who can understand the test instructions. It will be conducted on a cycle ergometer (Schiller 2000) using a ramp protocol tailored to each subject. After the test, acquired resting and peak exercise parameters will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) after Fontan operation

Exclusion Criteria:

* Active protein losing enteropathy
* Disability preventing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will invite adult patients who have undergone Fontan surgery and are followed up in the Adult Congenital Heart Disease Clinic at the Clinical Department of Cardiology, University Medical Centre Ljubljana. Patients with a known protein-losing enteropathy following Fontan surgery will be excluded. The control group will consist of patients who have undergone surgical or percutaneous repair of simple congenital heart defects (atrial or ventricular septal defects) without clinical signs of heart failure and with normal systemic venous pressure as assessed by ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Serum biomarkers of intestinal barrier dysfunction | Baseline
  Patients after Fontan operation will have higher serum biomarkers of intestinal barrier dysfunction in comparison to the control group
Serum biomarkers of systemic inflammation | Baseline
  Patients after Fontan operation will have higher serum biomarkers of systemic inflammatory response in comparison to the control group
Assessment of nutritional disorders | Baseline
  Patients after Fontan operation will have more nutritional disorders in comparison to the control group

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Pavšič, MD, PhD, Principal Investigator — UMC Ljubljana, Slovenia
Locations (1):
- University medical centre Ljubljana (UKC Ljubljana), Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
We will individually assess all requests for IPD.

REFERENCES:
- [Background] Go K, Horiba K, Yamamoto H, Morimoto Y, Fukasawa Y, Ohashi N, Yasuda K, Ishikawa Y, Kuraishi K, Suzuki K, Ito Y, Takahashi Y, Kato T. Dysbiosis of gut microbiota in patients with protein-losing enteropathy after the Fontan procedure. Int J Cardiol. 2024 Feb 1;396:131554. doi: 10.1016/j.ijcard.2023.131554. Epub 2023 Oct 22. PMID 37875211
- [Background] Saraf A, De Staercke C, Everitt I, Haouzi A, Ko YA, Jennings S, Kim JH, Rodriguez FH, Kalogeropoulos AP, Quyyumi A, Book W. Biomarker profile in stable Fontan patients. Int J Cardiol. 2020 Apr 15;305:56-62. doi: 10.1016/j.ijcard.2020.01.012. Epub 2020 Jan 9. PMID 31959411
- [Background] Sharma R, Bolger AP, Li W, Davlouros PA, Volk HD, Poole-Wilson PA, Coats AJ, Gatzoulis MA, Anker SD. Elevated circulating levels of inflammatory cytokines and bacterial endotoxin in adults with congenital heart disease. Am J Cardiol. 2003 Jul 15;92(2):188-93. doi: 10.1016/s0002-9149(03)00536-8. PMID 12860222
- [Background] Rychik J, Atz AM, Celermajer DS, Deal BJ, Gatzoulis MA, Gewillig MH, Hsia TY, Hsu DT, Kovacs AH, McCrindle BW, Newburger JW, Pike NA, Rodefeld M, Rosenthal DN, Schumacher KR, Marino BS, Stout K, Veldtman G, Younoszai AK, d'Udekem Y; American Heart Association Council on Cardiovascular Disease in the Young and Council on Cardiovascular and Stroke Nursing. Evaluation and Management of the Child and Adult With Fontan Circulation: A Scientific Statement From the American Heart Association. Circulation. 2019 Aug 6;140(6):e234-e284. doi: 10.1161/CIR.0000000000000696. Epub 2019 Jul 1. PMID 31256636
- [Background] Valentova M, von Haehling S, Bauditz J, Doehner W, Ebner N, Bekfani T, Elsner S, Sliziuk V, Scherbakov N, Murin J, Anker SD, Sandek A. Intestinal congestion and right ventricular dysfunction: a link with appetite loss, inflammation, and cachexia in chronic heart failure. Eur Heart J. 2016 Jun 1;37(21):1684-91. doi: 10.1093/eurheartj/ehw008. Epub 2016 Feb 9. PMID 26865478